CLINICAL TRIAL: NCT02562807
Title: A Phase I Study of TAS-303 in Female Patients With Stress Urinary Incontinence
Brief Title: A Study of TAS-303 in Female Patients With Stress Urinary Incontinence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10060040
Record Dates: First submitted 2015-09-18; First posted 2015-09-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Lower Urinary Tract Symptoms | interventions — TAS-303

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): TAS-303 18mg single-dose and then Placebo single-dose.
  Interventions: Drug: TAS-303 18mg single-dose; Drug: Placebo 18mg single-dose
- Treatment B (Placebo Comparator): Placebo single-dose and then TAS-303 18mg single-dose.
  Interventions: Drug: TAS-303 18mg single-dose; Drug: Placebo 18mg single-dose
- Treatment C (Active Comparator): TAS-303 9mg single-dose and then Placebo single-dose.
  Interventions: Drug: TAS-303 9mg single-dose; Drug: Placebo 9mg single-dose
- Treatment D (Placebo Comparator): TAS-303 Placebo single-dose and then TAS-303 9mg single-dose.
  Interventions: Drug: TAS-303 9mg single-dose; Drug: Placebo 9mg single-dose

INTERVENTIONS:
Drug: TAS-303 18mg single-dose
  Arms: Treatment A; Treatment B
Drug: Placebo 18mg single-dose
  Arms: Treatment A; Treatment B
Drug: TAS-303 9mg single-dose
  Arms: Treatment C; Treatment D
Drug: Placebo 9mg single-dose
  Arms: Treatment C; Treatment D

SUMMARY:
The purpose of this study is to evaluate pharmacological effect, safety and pharmacokinetic of TAS-303 in female patients with Stress Urinary Incontinence.

DETAILED DESCRIPTION:
This study is double-blind, placebo-controlled crossover study. The main purpose of this study is to evaluate Urethral Pressure Profile Parameters in Stress Urinary Incontinence patients who will receive single dose of TAS-303 or Placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has symptoms of Stress Urinary Incontinence (SUI) for at least 12 weeks prior to study entry
* Patient weights at least 45 kg and has body mass index (BMI) range of 18.0-30.0 kg/m2, inclusive, at screening
* Patient is positive in 1-hour pad weight test at screening
* Patient has at least 2 incontinence episodes per week.

Key Exclusion Criteria:

* Patient has predominant or primary urge incontinence according to investigator judgment
* Patient had a prior surgical SUI treatment
* Patient is diagnosed Pelvic Organ Prolapse
* Patient is currently taking medication, or has taken medication in the last 4 weeks, for urinary incontinence or that effect urinary output function including anti-cholinergic or anti-histamines or any anti-anxiety medications.
* Patient is positive pregnancy test

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Maximum Urethral Closure Pressure (MUCP) | Baseline, 6 hours after the administration

SECONDARY OUTCOMES:
Urethral pressure profile parameters: mean urethral closure pressure, functional profile length | Baseline, 6 hours after the administration
Safety assessed by incidence and severity of adverse events | Up to 36 days after the administration
Maximum plasma concentration (Cmax) of TAS-303 | 1, 2, 4, 6, 8, 12, 24, 48, 72 hours after the administration
Time to maximum plasma concentration (tmax) of TAS-303 | 1, 2, 4, 6, 8, 12, 24, 48, 72 hours after the administration
Area under the plasma concentration versus time curve (AUC) of TAS-303 | Immediately prior to dosing, and 1, 2, 4, 6, 8, 12, 24, 48, 72 hours after the administration
Elimination half-time (t1/2) of TAS-303 | 1, 2, 4, 6, 8, 12, 24, 48, 72 hours after the administration

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- Taiho Pharmaceutical Co., Ltd selected site, Kumamoto, Japan